CLINICAL TRIAL: NCT02571920
Title: Hemodynamic Monitoring, Positive Inotropic and Vasoactive Drugs During Cardiac Surgery (EMOA Study)
Brief Title: Hemodynamic Monitoring, Positive Inotropic and Vasoactive Drugs During Cardiac Surgery (EMOA)
Acronym: EMOA
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A14-D64-VOL.23
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: cardiac surgery; cardiac output

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Describe the proportion of patients who underwent cardiac surgery in France and benefiting from a monitoring cardiac output, describe the use of positive inotropic and vasoactive agents for cardiac surgery patients operated (type of catecholamines, their duration), describe the fluid replacement and transfusions of first 24 hours, describe the incidence of postoperative complications in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
The perioperative management in cardiac surgery patients has changed dramatically in the last fifteen years with the development of new cardiac output monitoring devices, the availability of new inotropic molecules, and a modern treatment for cardio-circulatory failure.

However, few studies report the possible changes in practice. The last French national survey was conducted in 2001. Since then, the literature is poor on the subject, and the impact of new approaches has been only marginally addressed. Recently, a German postal survey was conducted among cardiac surgery anesthesiologists, but on purely declarative elements and without patient data.

The investigators offer a type of national prospective observational study to evaluate professional practices, morbidity and mortality in cardiac surgical patients. This study must include all patients undergoing cardiac surgery at the participating centers during 7 weeks.

The main objective of this work is to assess the proportion of patients undergoing cardiac surgery receiving a cardiac output monitoring.

Secondary objectives are to describe the relationship between the use of cardiac output monitoring and the use of positive inotropic agents and vasoactive (type molecules, duration), volume expansion and transfusions the first 24 hours, and the incidence postoperative complications for patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old undergoing cardiac surgery during the study period

Non-inclusion Criteria:

* age under 18 years old
* Extracorporeal life support and others cardiac assistance
* congenital cardiac surgery
* TAVI procedures
* Pericardium surgical drainages
* Sternal sepsis surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving elective cardiac surgery during the study period
Sampling Method: Non-Probability Sample
Enrollment: 3099 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients undergoing cardiac surgery and receiving a cardiac output monitoring. | Up to 28 days after surgery (length of intensive care unit stay)

SECONDARY OUTCOMES:
Correlation between use of cardiac output monitoring and the incidence of norepinephrine use | Up to 28 days after surgery (length of intensive care unit stay)
Correlation between use of cardiac output monitoring and the incidence of dobutamine use | Up to 28 days after surgery (length of intensive care unit stay)
Correlation between use of cardiac output monitoring and the incidence of epinephrine use | Up to 28 days after surgery (length of intensive care unit stay)
Correlation between use of cardiac output monitoring and the length of norepinephrine infusion | Up to 28 days after surgery (length of intensive care unit stay)
Correlation between use of cardiac output monitoring and the length of dobutamine infusion | Up to 28 days after surgery (length of intensive care unit stay)
Correlation between use of cardiac output monitoring and the length of epinephrine infusion | Up to 28 days after surgery (length of intensive care unit stay)
Correlation between use of of cardiac output monitoring and the incidence of red blood cell transfusion | Up to 28 days after surgery (length of intensive care unit stay)
Correlation between use of of cardiac output monitoring and the volume of fluid expansion during first day following cardiac surgery | Up to 28 days after surgery (length of intensive care unit stay)
Correlation between use of of cardiac output monitoring and the incidence of postoperative complications | Up to 28 days after surgery (length of intensive care unit stay)

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Olivier Fischer, Principal Investigator — University Hospital, Caen; Fabien Dechanet, Principal Investigator — University Hospital, Caen; Raphaël D'Orlando, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France